CLINICAL TRIAL: NCT00846846
Title: Patient Related OuTcomes With Endeavor Versus Cypher Stenting Trial: PROTECT Continued Access Post Marketing Surveillance Trial
Brief Title: PROTECT Continued Access Post Marketing Surveillance Trial
Acronym: PROTECT-CA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medtronic Vascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Version 1.0, 29 October 2008
Record Dates: First submitted 2009-02-18; First posted 2009-02-19 (Estimated); Results first posted 2014-07-02 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-04

CONDITIONS: Coronary Artery Disease, Autosomal Dominant, 1
MeSH Terms: conditions — Coronary Artery Disease, Autosomal Dominant, 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Endeavor® Zotarolimus Eluting Coronary Stent (Experimental): Endeavor® Zotarolimus Eluting Coronary Stent System
  Interventions: Device: Endeavor® Zotarolimus Eluting Coronary Stent System

INTERVENTIONS:
Device: Endeavor® Zotarolimus Eluting Coronary Stent System — Endeavor® Zotarolimus Eluting Coronary Stent System in a patient population requiring stent implantation

SUMMARY:
In order to expand safety information in patients treated with the Endeavor Drug Eluting Stent System, or next generation model, a Continued Access (CA) study is added to the PROTECT Trial. The amended study is "PROTECT CONTINUED ACCESS" ("PROTECT CA").

DETAILED DESCRIPTION:
This was a prospective, multicenter, non-randomized, single-arm, open-label post market surveillance study designed to expand safety information in patients treated with the Endeavor® Zotarolimus Eluting Coronary Stent System.

Since their introduction, Drug Eluting Stents (DES) have markedly decreased stent restenosis and the clinical need for repeat revascularization frequently observed with bare metal stents (BMS)1-10. However, the widespread use of DES has raised concerns regarding the occurrence of late stent thrombosis (> 30 days after stent implantation)12-14. Although the incidence might seem low (0.2-0.7%)13,15-18 the high mortality and morbidity associated with stent thrombosis, and the soaring number of stents implanted annually, make it a significant medical problem.

The purpose of this trial was to investigate the long-term clinical safety and efficacy of the Endeavor drug eluting stent in a large and higher risk patient population, which more closely reflects clinical practice today. Both unstable and stable patients with single or multivessel disease and complex lesions were eligible for enrollment.

The selected primary endpoint was stent thrombosis, defined as definite and probable stent thrombosis according to the ARC definition, at 3 years. The main secondary endpoints were the composite of death or cardiac death combined with large or all non-fatal myocardial infarction, which are the typical clinical manifestations of stent thrombosis. These events are adjudicated by a clinical events committee.

1.2 Study Endpoints 1.2.1 Primary Endpoint: The overall stent thrombosis rate defined as definite and probable stent thrombosis according to the ARC definition at 3 years 1.2.2 Secondary Endpoints:

Main Secondary Endpoints include:

* Composite endpoint of total death and number of patients with all non-fatal myocardial infarction at 3 years
* Composite endpoint of cardiac death and number of patients with all non-fatal myocardial infarction at 3 years
* Composite endpoint of total death and number of patients with large non-fatal myocardial infarction at 3 years
* Composite endpoint of cardiac death and number of patients with large non-fatal myocardial infarction at 3 years

Additional secondary endpoints include:

* Total Death and subcategories of Death
* Large and all Myocardial Infarction (MI)
* Stent thrombosis defined as definite, probable and possible
* Composite score of clinical outcomes (death, myocardial infarction, stroke and revascularization) *
* Major Adverse Cardiac and Cerebral Events (MACCE)
* Stroke (hemorrhagic in nature while on clopidogrel)
* Bleeding complications in general
* Target lesion revascularization (TLR)
* Target vessel revascularization (TVR)
* Non target vessel revascularization (non TVR)
* Procedural success
* Device success
* Lesion success
* Endpoints will be calculated at the follow-up time points and for the mean follow-up period.

  * The composite score of clinical outcomes (death, myocardial infarction, stroke and revascularization) constructed from a patient population according to the Delphi method.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is > 18 years of age (or minimum age as required by local regulations).
2. The patient or patient's legal representative has consented to participate and has authorized the collection and release of his medical information by signing the "Patient Informed Consent Form".
3. All lesions requiring interventions (target lesions - one to a maximum of four) in one or more native coronary arteries are amendable for implantation of one or more Endeavor® Zotarolimus Eluting Coronary Stent System.
4. Patient indication, lesion length and vessel diameter of the target lesion(s) are according to the 'Indications for Use' as mentioned in the 'Instructions for Use' that comes with every Endeavor® Zotarolimus Eluting Coronary Stent System. Please check the 'Instructions for Use' that comes with the product. Please be aware that the 'Instructions for Use' may be subject to change during the course of the study.

5 The patient is willing and able to cooperate with study procedures and required follow up visits.

Exclusion Criteria:

1. Women with known pregnancy or who are lactating.
2. Planned elective surgery necessitating discontinuation of clopidogrel within the regular planned period of clopidogrel administration.
3. Patients expected not to be compliant with the anti-platelet and/or anticoagulation therapy regimen.
4. Previous brachytherapy.
5. Previous implantation of a drug eluting stent.
6. Previous implantation of a bare metal stent in the preceding year.
7. Simultaneous or planned intervention other non cardiac vessels including but not limited to renal artery or carotid artery.
8. Current medical condition with a life expectancy of less than 3 years.
9. Manifest acute severe heart failure (Killip class III-IV).
10. The patient is currently, and during the first 3 years of the PROTECT trial, participating in another investigational device or drug study that clinically interferes with the PROTECT-study endpoints; or requires coronary angiography or other coronary artery imaging procedures. The patient may only be enrolled in the PROTECT-study once.
11. Patients with medical conditions that preclude the follow-up as defined in the protocol or that otherwise limits participation in this study.
12. Patients on warfarin or similar anti-coagulant therapy.
13. Patients with hypersensitivity or allergies to one of the drugs or components indicated in the Instructions for Use.
14. Patients who are judged to have a lesion that prevents complete inflation of an angioplasty balloon.
15. Patients in whom anti-platelet and/or anticoagulation therapy is contraindicated.

16 Transplant patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1018 (Actual)
Dates: Start 2009-01; Primary Completion 2013-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Bousquette, Study Director — Medtronic Cardiovascular
Locations (1):
- University of Massachusetts Memorial Medical Center, Worcester, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1018 patients were enrolled from February 2009 until November 2009 in 48 participating hospitals in USA.
Pre-assignment Details: Subjects were excluded from participation if they did not meet inclusion/exclusion criteria.
Groups:
- Endeavor® Zotarolimus Eluting Coronary Stent System: Endeavor® Zotarolimus Eluting Coronary Stent System>
  > Endeavor® Zotarolimus Eluting Coronary Stent System: Endeavor® Zotarolimus Eluting Coronary Stent System in a patient population requiring stent implantation
Period: Overall Study
Arm/Group | Endeavor® Zotarolimus Eluting Coronary Stent System
Started | 1018
Completed | 943 (Study ongoing but not recruiting participants.)
Not Completed | 75
Not completed — Death | 56
Not completed — Withdrawal by Subject | 19

BASELINE CHARACTERISTICS:
Groups:
- Endeavor® Zotarolimus Eluting Coronary Stent System: Endeavor® Zotarolimus Eluting Coronary Stent Implantation in a patient population requiring stent implantation.
Arm/Group | Endeavor® Zotarolimus Eluting Coronary Stent System
Number analyzed (Participants) | 1018
Age, Continuous [Mean (Full Range); unit: Years] | 63.16 [31 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 274
  Male | 744
Region of Enrollment [Number; unit: participants]
  United States | 1018

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate Overall Stent Thrombosis Rate of the Endeavor® Zotarolimus Eluting Coronary Stent System in a Patient Population Requiring Stent Implantation
Description: The primary endpoint rate of ARC-defined definite or probable stent thrombosis at 3 years.
Time Frame: 3 years
Population: Of the one thousand and eighteen (1018) ITT patients, a total of nine hundred and forty seven (947) patients were included in the primary endpoint analysis. These patients had at least 1050 days of follow-up or had experienced stent thrombosis prior to 1080 days.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Endeavor® Zotarolimus Eluting Coronary Stent System: Intention to treat analyis has been used.
Arm/Group | Endeavor® Zotarolimus Eluting Coronary Stent System
Number analyzed (Participants) | 947
percentage of participants | 1.2 [0.6 to 2.1]

2. Secondary Outcome: Composites of (Cardiac) Death and (Large) Non-fatal Myocardial Infarctions.
Description: Total death and and number of patients with all non-fatal myocardial infarction. Cardiac death and number of patients with all non-fatal myocardial infarction. Total death and number of patients with large non-fatal myocardial infarction. Cardiac death and number of patients with large non-fatal myocardial infarction.
Time Frame: 3 years
Population: Main secondary endpoint results for the ITT population are similar to the primary endpoint analysis, a total of nine hundred and forty seven (947) ITT patients had sufficient follow-up or an event to be included in the main secondary endpoint analyses.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Endeavor® Zotarolimus Eluting Coronary Stent System
Number analyzed (Participants) | 947
percentage of participants
  the composite rate of death and/or MI | 11.7 [9.7 to 13.9]
  the composite rate of cardiac death and/or MI | 8.2 [6.6 to 10.2]
  composite rate of death and/or large MI | 7.8 [6.2 to 9.7]
  composite rate of cardiac death and/or large MI | 4.2 [3.0 to 5.7]

ADVERSE EVENTS:
Time Frame: 12 months
Groups:
- Endeavor: Medtronic Endeavor
Arm/Group | Endeavor
Serious Adverse Events (participants affected / at risk) | 415/1018
Other Adverse Events (participants affected / at risk) | 134/1018
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Endeavor (N=1018)
Anaemia (Blood and lymphatic system disorders) | 10 (12)
Acute Myocardial Infarction (Cardiac disorders) | 30 (36)
Angina Pectoris (Cardiac disorders) | 49 (55)
Angina Unstable (Cardiac disorders) | 26 (31)
Atrial Fibrillation (Cardiac disorders) | 16 (19)
Bradycardia (Cardiac disorders) | 7 (7)
Cardiac Failure Congestive (Cardiac disorders) | 12 (25)
Cardiac Tamponade (Cardiac disorders) | 1 (1)
Cardiogenic Shock (Cardiac disorders) | 3 (3)
Coronary Artery Disease (Cardiac disorders) | 22 (25)
Coronary Artery Dissection (Cardiac disorders) | 28 (29)
Coronary Artery Occlusion (Cardiac disorders) | 2 (2)
Coronary Artery Restenosis (Cardiac disorders) | 5 (5)
Coronary Artery Stenosis (Cardiac disorders) | 5 (5)
In-Stent Coronary Artery Restenosis (Cardiac disorders) | 17 (18)
Myocardial Infarction (Cardiac disorders) | 17 (17)
Pericarditis (Cardiac disorders) | 1 (1)
Supraventricular Tachycardia (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 2 (2)
Ventricular Fibrillation (Cardiac disorders) | 2 (2)
Ventricular Tachycardia (Cardiac disorders) | 4 (4)
Vertigo (Ear and labyrinth disorders) | 3 (3)
Abdominal Pain (Gastrointestinal disorders) | 14 (15)
Diarrhoea (Gastrointestinal disorders) | 5 (5)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 24 (28)
Gastrointestinal Ulcer (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2)
Chest Discomfort (General disorders) | 9 (9)
Chest Pain (General disorders) | 69 (93)
Death (General disorders) | 6 (6)
Fatigue (General disorders) | 1 (1)
Hernia (General disorders) | 3 (3)
Non-Cardiac Chest Pain (General disorders) | 12 (13)
Oedema Peripheral (General disorders) | 2 (2)
Pyrexia (General disorders) | 1 (1)
Unevaluable Event (General disorders) | 151 (237)
Vessel Puncture Site Haematoma (General disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 3 (3)
Bronchitis (Infections and infestations) | 9 (10)
Diverticulitis (Infections and infestations) | 2 (3)
Infection (Infections and infestations) | 4 (4)
Pneumonia (Infections and infestations) | 17 (20)
Urinary Tract Infection (Infections and infestations) | 5 (8)
Stent Occlusion (Injury, poisoning and procedural complications) | 2 (2)
Thrombosis In Device (Injury, poisoning and procedural complications) | 9 (9)
Cardiac Enzymes Increased (Investigations) | 9 (9)
Electrocardiogram ST Segment Elevation (Investigations) | 1 (1)
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 (1)
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 9 (9)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 7 (8)
Cerebrovascular Accident (Nervous system disorders) | 22 (23)
Dizziness (Nervous system disorders) | 2 (2)
Presyncope (Nervous system disorders) | 2 (2)
Syncope (Nervous system disorders) | 11 (12)
Transient Ischaemic Attack (Nervous system disorders) | 5 (5)
Depression (Psychiatric disorders) | 2 (2)
Haematuria (Renal and urinary disorders) | 6 (8)
Renal Failure (Renal and urinary disorders) | 11 (11)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 21 (23)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Arterial Occlusive Disease (Vascular disorders) | 1 (1)
Arteriovenous Fistula (Vascular disorders) | 1 (1)
Haematoma (Vascular disorders) | 2 (2)
Haemorrhage (Vascular disorders) | 7 (8)
Hypertension (Vascular disorders) | 5 (6)
Hypotension (Vascular disorders) | 5 (6)
Peripheral Ischaemia (Vascular disorders) | 2 (2)
Vascular Pseudoaneurysm (Vascular disorders) | 4 (4)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Endeavor (N=1018)
Unevaluable Event (General disorders) | 134 (190)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For any publication or presentation of the Protected Materials or any portion thereof, a maunscript of the paper, abstract or any materials will be provided by Consultant to Sponsor for its approval at least sixty (60days) for manuscripts and thirty (30) days for presentations prior to outside submission. Medtronic shall have the right to request reasonable modifications of any manuscript or other materials to be published or presented.